CLINICAL TRIAL: NCT00224874
Title: Initial Systemic Treatment of Acute GVHD: A Phase II Randomized Trial Evaluating Etanercept, Mycophenolate Mofetil (MMF), Denileukin Diftitox (ONTAK), and Pentostatin in Combination With Corticosteroids (BMT CTN #0302)
Brief Title: Treatment for Acute Graft-Versus-Host Disease (BMT CTN 0302)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH); Blood and Marrow Transplant Clinical Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMTCTN0302; BMT CTN 0302 (Other: Blood and Marrow Transplant Clinicial Trials Network); U01HL069294-05 (NIH); 285 (Other: National Heart, Lung, and Blood Institute); NCT00253656 (obsolete NCT alias); NCT00474149 (obsolete NCT alias)
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Results first posted 2010-04-09 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2017-08

CONDITIONS: Graft vs Host Disease; Immune System Disorders
Keywords: Acute Graft vs Host Disease; GVHD
MeSH Terms: conditions — Graft vs Host Disease; Immune System Diseases | interventions — Etanercept; Mycophenolic Acid; denileukin diftitox; Pentostatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Etanercept (Experimental): Enroll within 48 hours of new onset acute GVHD and randomize to Etanercept
  Interventions: Drug: Etanercept
- Mycophenolate Mofetil (Experimental): Enroll within 48 hours of new onset acute GVHD and randomize to Mycophenolate Mofetil
  Interventions: Drug: Mycophenolate Mofetil
- Denileukin Diftitox (Experimental): Enroll within 48 hours of new onset acute GVHD and randomize to Denileukin Diftitox
  Interventions: Drug: Denileukin Diftitox
- Pentostatin (Experimental): Enroll within 48 hours of new onset acute GVHD and randomize to Pentostatin
  Interventions: Drug: Pentostatin

INTERVENTIONS:
Drug: Etanercept — Etanercept [25 mg subcutaneously twice weekly for up to 4 weeks; discontinue if in complete response by 4 weeks].
  Other Names: ENBREL®
  Arms: Etanercept
Drug: Mycophenolate Mofetil — Mycophenolate mofetil (MMF) [20 mg/kg (maximum 1 gm) orally or intravenously twice daily; continue through prednisone taper, then taper MMF over 4 weeks].
  Other Names: CellCept®
  Arms: Mycophenolate Mofetil
Drug: Denileukin Diftitox — Denileukin Diftitox (ONTAK®) [9 mcg/kg intravenously Days 1, 3, 5, 15, 17, 19].
  Other Names: ONTAK®
  Arms: Denileukin Diftitox
Drug: Pentostatin — Pentostatin [1.5 mg/m2 daily for 3 days; Days 1-3 and repeat Days 15-17
  Other Names: Nipent®
  Arms: Pentostatin

SUMMARY:
The study is a randomized Phase II, four arm treatment trial. The primary purpose of the study is to define new agents with promising activity against acute graft-versus-host disease (GVHD) suitable for testing against corticosteroids alone in a subsequent Phase III trial.

DETAILED DESCRIPTION:
BACKGROUND:

Acute graft-versus-host disease (GVHD) is the major complication of allogeneic hematopoietic stem cell (HSC) transplantation. Acute GVHD produces significant morbidity and complicates patient management resulting in organ toxicity, frequent infections, malnutrition, and substantial delay in recovery from transplantation. Corticosteroids have been the primary therapy for acute GVHD for over three decades. Various additional immunosuppressive strategies have been tested as GVHD therapy but neither anti-thymocyte globulin (ATG), CD5-immunotoxins, IL-1 antagonists nor other agents have been demonstrably helpful in either control of GVHD symptoms or improvement in survival. Published response rates of complete response (CR) to acute GVHD therapy with corticosteroids range from 25-41%. These rates will be used as benchmarks for assessing efficacy of promising new agents. New immunosuppressive agents and strategies are required to improve the management of GVHD and decrease the toxicities of the immunosuppressive regimens.

DESIGN NARRATIVE:

In this trial, patients with newly diagnosed acute GVHD will be randomly assigned to receive corticosteroids plus one of four new agents (etanercept, MMF, denileukin diftitox [Ontak], and pentostatin). A control arm of only corticosteroids will not be employed. Each agent will be assessed for safety and efficacy (at least 35% complete remission [CR] rate at Day 28 of therapy can be expected from previously untreated patients).

ELIGIBILITY:
Inclusion Criteria:

* Prior allogeneic hematopoietic stem cell transplant using either bone marrow, peripheral blood stem cells, or cord blood
* De novo acute GVHD diagnosed within 48 hours prior to enrollment; biopsy confirmation of GVHD is strongly recommended but not required; enrollment should not be delayed awaiting biopsy or pathology results; the patient must have had no previous systemic immune suppressive therapy given for treatment of acute GVHD except for a maximum 48 hours of prior corticosteroid therapy (at least 1 mg/kg/day methylprednisolone)
* Patients that have undergone a scheduled donor lymphocyte infusion (DLI) as part of their original transplant therapy plan
* Absolute neutrophil count (ANC) greater than 500/µL
* Clinical status at enrollment to allow tapering of steroids to not less than 1 mg/kg/day methylprednisolone (1.4 mg/kg/day prednisone) at Day 28 of therapy (e.g., persisting malignant disease suggesting the need for accelerated taper of immunosuppression)
* Estimated creatinine clearance greater than 30 mL/minute
* Assent and educational materials provided to, and reviewed with, patients under the age of 18

Exclusion Criteria:

* ONTAK, pentostatin, or etanercept given within 7 days of enrollment
* Active uncontrolled infection
* Patients that have undergone an unscheduled DLI, or DLI that was not part of their original transplant therapy plan
* If any prior steroid therapy (for indication other than GVHD), treatment at doses of at least 0.5 mg/kg/day methylprednisolone within 7 days prior to onset of GVHD
* Patients unlikely to be available at the transplant center on Day 28 and 56 of therapy
* A clinical syndrome resembling de novo chronic GVHD developing at any time after allotransplantation (see Chapter 2 of the BMT CTN Manual of Procedures for details of de novo chronic GVHD)
* Other investigational therapeutics for GVHD within 30 days, including agents used for GVHD prophylaxis
* Patients who are pregnant, breast feeding, or if sexually active, unwilling to use effective birth control for the duration of the study
* Adults unable to provide informed consent
* Patients with a history of intolerance to any of the study drugs

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2005-09; Primary Completion 2009-01 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Horowitz, MD, Study Director — Center for International Blood and Marrow Transplant Research
Locations (19):
- United States (19):
  - City of Hope National Medical Center, Duarte, California
  - University of California, San Diego, California
  - Stanford Hospital and Clinics, Stanford, California
  - University of Florida College of Medicine (Shands), Gainesville, Florida
  - Johns Hopkins/SKCCC, Baltimore, Maryland
  - DFCI/Brigham & Women's Hospital, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University/Barnes Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke University Medical Center (Peds), Durham, North Carolina
  - University Hospitals of Cleveland/Case Western, Cleveland, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - University of Texas/MD Anderson CRC, Houston, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in a manuscript and supporting information submitted to NIH BioLINCC (including data dictionaries, case report forms, data submission documentation, documentation for outcomes dataset, etc where indicated).
Supporting Information: Study Protocol, ICF
Time Frame: Within 6 months of official study closure at participating sites.
Access Criteria: Available to the public
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Result] Alousi AM, Weisdorf DJ, Logan BR, Bolanos-Meade J, Carter S, Difronzo N, Pasquini M, Goldstein SC, Ho VT, Hayes-Lattin B, Wingard JR, Horowitz MM, Levine JE; Blood and Marrow Transplant Clinical Trials Network. Etanercept, mycophenolate, denileukin, or pentostatin plus corticosteroids for acute graft-versus-host disease: a randomized phase 2 trial from the Blood and Marrow Transplant Clinical Trials Network. Blood. 2009 Jul 16;114(3):511-7. doi: 10.1182/blood-2009-03-212290. Epub 2009 May 14. PMID 19443659
- [Result] Jacobson PA, Huang J, Wu J, Kim M, Logan B, Alousi A, Grimley M, Bolanos-Meade J, Ho V, Levine JE, Weisdorf D. Mycophenolate pharmacokinetics and association with response to acute graft-versus-host disease treatment from the Blood and Marrow Transplant Clinical Trials Network. Biol Blood Marrow Transplant. 2010 Mar;16(3):421-9. doi: 10.1016/j.bbmt.2009.11.010. PMID 19925875
- [Result] Levine JE, Logan B, Wu J, Alousi AM, Ho V, Bolanos-Meade J, Weisdorf D; Blood and Marrow Transplant Clinical Trials Network. Graft-versus-host disease treatment: predictors of survival. Biol Blood Marrow Transplant. 2010 Dec;16(12):1693-9. doi: 10.1016/j.bbmt.2010.05.019. Epub 2010 Jun 9. PMID 20541024
- [Derived] Levine JE, Logan BR, Wu J, Alousi AM, Bolanos-Meade J, Ferrara JL, Ho VT, Weisdorf DJ, Paczesny S. Acute graft-versus-host disease biomarkers measured during therapy can predict treatment outcomes: a Blood and Marrow Transplant Clinical Trials Network study. Blood. 2012 Apr 19;119(16):3854-60. doi: 10.1182/blood-2012-01-403063. Epub 2012 Mar 1. PMID 22383800

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Clinic patients were recruited from August 2005 through March 2008.
Groups:
- Etanercept: Patients received 25 mg Etanercept subcutaneously twice weekly for up to 4 weeks; discontinue if in Complete Response (CR) by 4 weeks
- Mycophenolate Mofetil: Patients received Mycophenolate Mofetil (MMF) 20 mg/kg (maximum 1 gm) per oral or intravenously twice daily; continue through prednisone taper, then taper MMF over 4 weeks
- Denileukin Diftitox: Patients received Denileukin Diftitox 9 mcg/kg intravenously over 1 hour on days 1, 3, 5, 15, 17, 19.
- Pentostatin: Patients received Pentostatin 1.5 mg/m2 intravenously daily on days 1-3 and 15-17.
Period: Overall Study
Arm/Group | Etanercept | Mycophenolate Mofetil | Denileukin Diftitox | Pentostatin
Started | 46 | 45 | 47 | 42
Completed | 46 | 45 | 46 | 42
Not Completed | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Etanercept | Mycophenolate Mofetil | Denileukin Diftitox | Pentostatin | Total
Number analyzed (Participants) | 46 | 45 | 47 | 42 | 180
Age, Continuous [Median (Full Range); unit: years] | 50 [8 to 70] | 42 [13 to 63] | 51 [11 to 67] | 53 [24 to 68] | 50 [8 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 19 | 15 | 67
  Male | 30 | 28 | 28 | 27 | 113
Primary Disease [Number; unit: participants]
  Acute Myeloid Leukemia (AML) / MDS | 24 | 21 | 24 | 20 | 89
  Acute Lymphoblastic Leukemia (ALL) | 6 | 9 | 4 | 7 | 26
  Chronic Myeloid Leukemia (CML) | 2 | 2 | 1 | 0 | 5
  Lymphoma | 5 | 6 | 8 | 6 | 25
  Other | 9 | 7 | 10 | 9 | 35
Conditioning Regimen [Number; unit: participants]
  Myeloablative | 29 | 37 | 25 | 26 | 117
  Non-myeloablative | 17 | 8 | 21 | 15 | 61
  Unknown | 0 | 0 | 1 | 1 | 2
Donor Status [Number; unit: participants]
  Related | 21 | 24 | 21 | 17 | 83
  Unrelated | 24 | 21 | 25 | 24 | 94
  Unknown | 1 | 0 | 1 | 1 | 3
Stem Cell Type [Number; unit: participants]
  Bone Marrow | 5 | 13 | 15 | 9 | 42
  Peripheral Blood | 36 | 29 | 19 | 27 | 111
  Umbilical Cord Blood | 5 | 3 | 12 | 5 | 25
  Unknown | 0 | 0 | 1 | 1 | 2
MMF Prophylaxis [Number; unit: participants]
  Yes | 14 | 0 | 16 | 14 | 44
  No | 32 | 45 | 31 | 28 | 136
Enrollment Acute GVHD [Number; unit: participants]
  Grade 0 | 1 | 0 | 0 | 0 | 1
  Grade I | 8 | 3 | 8 | 4 | 23
  Grade II | 25 | 25 | 23 | 26 | 99
  Grade III | 12 | 16 | 15 | 11 | 54
  Grade IV | 0 | 1 | 1 | 1 | 3
Organ Involvement at Randomization [Number; unit: participants] — Some participants had multiple organ involvement at time of randomization and are be considered in more then one category.
  participants
    Skin | 36 | 35 | 35 | 34 | 140
    GI tract, lower | 12 | 18 | 14 | 17 | 61
    GI tract, upper | 10 | 12 | 14 | 13 | 49
    Liver | 6 | 7 | 7 | 5 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Complete Response (CR) at Day 28 of Therapy
Description: Complete response at day 28 after randomization. CR was defined as resolution of all signs and symptoms of Graft-Versus-Host Disease (GVHD) in all evaluable organs in comparison to Day 1 scoring.
Time Frame: Measured at Day 28
Population: All patients randomized were included in the analysis on an intent-to-treat basis
Measure: Number; unit: participants
Arm/Group | Etanercept | Mycophenolate Mofetil | Denileukin Diftitox | Pentostatin
Number analyzed (Participants) | 46 | 45 | 47 | 42
participants | 12 | 27 | 25 | 16

2. Secondary Outcome: Number of Partial Response (PR), Mixed Response (MR), and Progression
Description: Partial response, mixed response, and progression at Day 28 after randomization. Partial response was defined as improvement in one or more organs involved with Graft-Versus-Host Disease (GVHD) symptoms without progression in others. Mixed response was defined as improvement in one or more organs with deterioration in another organ manifesting symptoms of GVHD or development of symptoms of GVHD in a new organ. Progression was defined as deterioration in at least one organ without any improvement in others.
Time Frame: Measured at Day 28
Population: All patients randomized were included in the analysis on an intent-to-treat basis
Measure: Number; unit: participants
Arm/Group | Etanercept | Mycophenolate Mofetil | Denileukin Diftitox | Pentostatin
Number analyzed (Participants) | 46 | 45 | 47 | 42
participants
  Partial Response | 10 | 8 | 3 | 10
  Mixed Response | 3 | 4 | 0 | 2
  Progression | 7 | 1 | 3 | 4

3. Secondary Outcome: Proportion of Treatment Failure
Time Frame: Measured at Day 56
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept | Mycophenolate Mofetil | Denileukin Diftitox | Pentostatin
Number analyzed (Participants) | 46 | 45 | 47 | 42
percentage of participants | 24 [12 to 36] | 9 [6 to 17] | 26 [13 to 38] | 29 [15 to 42]

4. Secondary Outcome: Number of Patients With Acute Graft-versus-host Disease (GVHD) Flares at Day 90
Description: Flares were defined as any increase in symptoms of or therapy for acute GVHD after an initial response (i.e., progression from an earlier CR or PR).
Time Frame: Measured at Day 90
Population: All patients randomized were included in the analysis on an intent-to-treat basis
Measure: Number; unit: participants
Arm/Group | Etanercept | Mycophenolate Mofetil | Denileukin Diftitox | Pentostatin
Number analyzed (Participants) | 46 | 45 | 47 | 42
participants | 16 [0.21 to 0.49] | 12 [0.14 to 0.40] | 15 [0.21 to 0.49] | 15 [0.21 to 0.50]

5. Secondary Outcome: Number of Patients Discontinuing Immune Suppression Without Flare
Description: Immunosuppression discontinuation was defined as the discontinuation of corticosteroids and all additional immunosuppressives, except cyclosporine or tacrolimus, for treatment of acute GVHD without subsequent flare by Day 90 post-initiation of therapy and later by discontinuation of all immunosuppressive medications, including cyclosporine or tacrolimus.
Time Frame: Measured at Days 90, 180, and 270 post-treatment
Population: All patients randomized were included in the analysis on an intent-to-treat basis
Measure: Number; unit: participants
Arm/Group | Etanercept | Mycophenolate Mofetil | Denileukin Diftitox | Pentostatin
Number analyzed (Participants) | 46 | 45 | 47 | 42
participants
  Day 90 | 7 [0.05 to 0.26] | 4 [0.01 to 0.17] | 5 [0.02 to 0.19] | 2 [0 to 0.11]
  Day 180 | 12 [0.13 to 0.39] | 13 [0.16 to 0.42] | 8 [0.06 to 0.28] | 8 [0.07 to 0.31]
  Day 270 | 16 [0.21 to 0.49] | 17 [0.24 to 0.52] | 10 [0.10 to 0.33] | 10 [0.11 to 0.37]

6. Secondary Outcome: Number of Patients With Chronic Graft-versus-host Disease (GVHD)
Description: Number of patients with limited and extensive chronic GVHD at 9 months
Time Frame: Measured at 9 months
Population: All patients randomized were included in the analysis on an intent-to-treat basis
Measure: Number; unit: participants
Arm/Group | Etanercept | Mycophenolate Mofetil | Denileukin Diftitox | Pentostatin
Number analyzed (Participants) | 46 | 45 | 47 | 42
participants | 11 | 19 | 15 | 12

7. Secondary Outcome: Number of Patients Surviving at 6 and 9 Months Post Randomization
Time Frame: Measured at 6 and 9 months
Population: All patients randomized were included in the analysis on an intent-to-treat basis
Measure: Number; unit: participants
Arm/Group | Etanercept | Mycophenolate Mofetil | Denileukin Diftitox | Pentostatin
Number analyzed (Participants) | 46 | 45 | 47 | 42
participants
  Month 6 | 26 [0.43 to 0.72] | 32 [0.54 to 0.82] | 28 [0.47 to 0.76] | 24 [0.38 to 0.69]
  Month 9 | 22 [0.32 to 0.61] | 29 [0.48 to 0.76] | 24 [0.34 to 0.62] | 21 [0.31 to 0.62]

8. Secondary Outcome: Cumulative Incidence of Systemic Infections
Time Frame: Measured at Day 270
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept | Mycophenolate Mofetil | Denileukin Diftitox | Pentostatin
Number analyzed (Participants) | 46 | 45 | 47 | 42
percentage of participants | 47 [33 to 63] | 44 [30 to 59] | 62 [48 to 76] | 57 [42 to 72]

9. Secondary Outcome: Incidence of Epstein-Barr Virus (EBV)-Associated Lymphoma
Time Frame: Measured at 9 months
Population: No data collected
Arm/Group | Etanercept | Mycophenolate Mofetil | Denileukin Diftitox | Pentostatin
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Start of study through 9 months after randomization.
Description: Unexpected Adverse Events Included
Arm/Group | Etanercept | Mycophenolate Mofetil | Denileukin Diftitox | Pentostatin
Serious Adverse Events (participants affected / at risk) | 4/46 | 2/45 | 2/47 | 7/42
Other Adverse Events (participants affected / at risk) | 0/46 | 0/45 | 0/47 | 0/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=46) | Mycophenolate Mofetil (N=45) | Denileukin Diftitox (N=47) | Pentostatin (N=42)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Adverse drug reaction (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2007-08-20): https://cdn.clinicaltrials.gov/large-docs/74/NCT00224874/Prot_SAP_ICF_000.pdf